CLINICAL TRIAL: NCT00986648
Title: A Multi-Center Group to Study Acute Liver Failure in Children
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1U01DK072146-01 (NIH); U01DK072146 (NIH); 2U01DK072146-06 (NIH)
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Acute Liver Failure; Hepatic Encephalopathy
Keywords: acute liver failure; hepatic encephalopathy; acetaminophen toxicity
MeSH Terms: conditions — Liver Failure, Acute; Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The PALF study group began with 20 sites and now continues with 12 sites (11 in the United States and 1 in Canada) in the new funding period. The primary objective of the Pediatric Acute Liver Failure (PALF) study is to collect, maintain, analyze, and report clinical, epidemiological, and outcome data in children with ALF, including information derived from biospecimens.

DETAILED DESCRIPTION:
The PALF study group will collect clinical, epidemiological and outcome data on children with ALF. This information will be used to develop methods to predict whether a child will recover from the illness without the need for a liver transplant or other life-saving procedure. We believe the methods to predict survival will vary with different patient age groups, but that diagnosis, multi-system organ failure, degree of encephalopathy and level of coagulopathy will be important regardless of patient age. Biological samples, such as blood and liver tissue, will provide opportunities to identify subgroups of patients who have unique treatment requirements and outcomes. In addition, we hope to identify unrecognized mechanisms of liver injury resulting in ALF in children. Eligible study participants will be invited to participate in neurocognitive testing. Since patients that develop acute liver failure experience varying levels of hepatic encephalopathy and cerebral edema, we suspect that there may be residual sub-clinical neurological injury that compromises long-term neurocognitive function. Detailed neurocognitive testing has never been performed in a cohort of children that survive acute liver failure and this study seeks to close that information gap by defining the spectrum of neurocognitive outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent
* Birth through 17 years of age
* Biochemical evidence of acute liver injury
* Coagulopathy not corrected by vitamin K (or other intervention intended to correct coagulopathy)

  * The presence of encephalopathy (ENC) is required if the INR is at least 1.5 and less than 2.0
  * If INR is at least 2.0, the presence of ENC is not required

Exclusion Criteria:

* Known chronic underlying liver disease
* Multi-organ system failure following heart surgery or ECMO
* Solid organ or bone marrow transplantation
* Acute trauma
* Previously enrolled in the PALF Cohort Study
* Other severe illness, condition, or other reason in the opinion of the investigator that would make the patient unsuitable for the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between birth and age 18 years who present with acute liver failure.
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2000-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Squires, MD, Principal Investigator — Children's Hospital of Pittsburgh of UPMC, University of Pittsburgh
Locations (20):
- United States (17):
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Emory University, Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard University, Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Columbia-Presbyterian, New York, New York
  - University of Cincinnati, Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - King's College Hospital (London, UK), London

REFERENCES:
- [Result] Narkewicz MR, Dell Olio D, Karpen SJ, Murray KF, Schwarz K, Yazigi N, Zhang S, Belle SH, Squires RH; Pediatric Acute Liver Failure Study Group. Pattern of diagnostic evaluation for the causes of pediatric acute liver failure: an opportunity for quality improvement. J Pediatr. 2009 Dec;155(6):801-806.e1. doi: 10.1016/j.jpeds.2009.06.005. Epub 2009 Jul 29. PMID 19643443
- [Result] Rudnick DA, Dietzen DJ, Turmelle YP, Shepherd R, Zhang S, Belle SH, Squires R; Pediatric Acute Liver Failure Study Group. Serum alpha-NH-butyric acid may predict spontaneous survival in pediatric acute liver failure. Pediatr Transplant. 2009 Mar;13(2):223-30. doi: 10.1111/j.1399-3046.2008.00998.x. Epub 2008 Jul 17. PMID 18643912
- [Result] James LP, Alonso EM, Hynan LS, Hinson JA, Davern TJ, Lee WM, Squires RH; Pediatric Acute Liver Failure Study Group. Detection of acetaminophen protein adducts in children with acute liver failure of indeterminate cause. Pediatrics. 2006 Sep;118(3):e676-81. doi: 10.1542/peds.2006-0069. PMID 16950959
- [Result] Squires RH Jr, Shneider BL, Bucuvalas J, Alonso E, Sokol RJ, Narkewicz MR, Dhawan A, Rosenthal P, Rodriguez-Baez N, Murray KF, Horslen S, Martin MG, Lopez MJ, Soriano H, McGuire BM, Jonas MM, Yazigi N, Shepherd RW, Schwarz K, Lobritto S, Thomas DW, Lavine JE, Karpen S, Ng V, Kelly D, Simonds N, Hynan LS. Acute liver failure in children: the first 348 patients in the pediatric acute liver failure study group. J Pediatr. 2006 May;148(5):652-658. doi: 10.1016/j.jpeds.2005.12.051. PMID 16737880
- [Result] Alonso EM. Acute liver failure in children: the role of defects in fatty acid oxidation. Hepatology. 2005 Apr;41(4):696-9. doi: 10.1002/hep.20680. No abstract available. PMID 15789368
- [Result] Shneider BL, Rinaldo P, Emre S, Bucuvalas J, Squires R, Narkewicz M, Gondolesi G, Magid M, Morotti R, Hynan LS. Abnormal concentrations of esterified carnitine in bile: a feature of pediatric acute liver failure with poor prognosis. Hepatology. 2005 Apr;41(4):717-21. doi: 10.1002/hep.20631. PMID 15791615
- [Result] Sundaram SS, Alonso EM, Narkewicz MR, Zhang S, Squires RH; Pediatric Acute Liver Failure Study Group. Characterization and outcomes of young infants with acute liver failure. J Pediatr. 2011 Nov;159(5):813-818.e1. doi: 10.1016/j.jpeds.2011.04.016. Epub 2011 May 31. PMID 21621221
- [Result] Sundaram V, Shneider BL, Dhawan A, Ng VL, Im K, Belle S, Squires RH. King's College Hospital Criteria for non-acetaminophen induced acute liver failure in an international cohort of children. J Pediatr. 2013 Feb;162(2):319-23.e1. doi: 10.1016/j.jpeds.2012.07.002. Epub 2012 Aug 18. PMID 22906509
- [Result] Leonis MA, Alonso EM, Im K, Belle SH, Squires RH; Pediatric Acute Liver Failure Study Group. Chronic acetaminophen exposure in pediatric acute liver failure. Pediatrics. 2013 Mar;131(3):e740-6. doi: 10.1542/peds.2011-3035. Epub 2013 Feb 25. PMID 23439908
- [Result] Bucuvalas J, Filipovich L, Yazigi N, Narkewicz MR, Ng V, Belle SH, Zhang S, Squires RH. Immunophenotype predicts outcome in pediatric acute liver failure. J Pediatr Gastroenterol Nutr. 2013 Mar;56(3):311-5. doi: 10.1097/MPG.0b013e31827a78b2. PMID 23111765
- [Result] Lu BR, Zhang S, Narkewicz MR, Belle SH, Squires RH, Sokol RJ; Pediatric Acute Liver Failure Study Group. Evaluation of the liver injury unit scoring system to predict survival in a multinational study of pediatric acute liver failure. J Pediatr. 2013 May;162(5):1010-6.e1-4. doi: 10.1016/j.jpeds.2012.11.021. Epub 2012 Dec 20. PMID 23260095
- [Derived] Feldman AG, Sokol RJ, Hardison RM, Alonso EM, Squires RH, Narkewicz MR; Pediatric Acute Liver Failure Study Group. Lactate and Lactate: Pyruvate Ratio in the Diagnosis and Outcomes of Pediatric Acute Liver Failure. J Pediatr. 2017 Mar;182:217-222.e3. doi: 10.1016/j.jpeds.2016.12.031. Epub 2017 Jan 12. PMID 28088395
- [Derived] Narkewicz MR, Horslen S, Belle SH, Rudnick DA, Ng VL, Rosenthal P, Romero R, Loomes KM, Zhang S, Hardison RM, Squires RH; Pediatric Acute Liver Failure Study Group. Prevalence and Significance of Autoantibodies in Children With Acute Liver Failure. J Pediatr Gastroenterol Nutr. 2017 Feb;64(2):210-217. doi: 10.1097/MPG.0000000000001363. PMID 27496798